CLINICAL TRIAL: NCT02704520
Title: Magnetic Resonance Tumour Regression Grade (mrTRG) as a Novel Biomarker to Stratify Management of Good and Poor Responders to Radiotherapy: A Rectal Cancer Multicentre Randomised Control Trial to Avoid Surgery With 'Watch and Wait' or Intensify Treatment According to mrTRG
Brief Title: Magnetic Resonance Tumour Regression Grade (mrTRG) as a Novel Biomarker - Phase III Non CTIMP Trial
Acronym: TRIGGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCUMAS: 23HH8209
Record Dates: First submitted 2016-02-05; First posted 2016-03-10 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Magnetic Resonance Imaging; Chemoradiotherapy; Chemotherapy; Diagnostic Imaging
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Other): Management according to national guidelines - conventional MDT, clinical assessment post-treatment planning
  Interventions: Diagnostic Test: High resolution MRI scan
- Intervention arm (Experimental): mrTRG directed management 'Good response' (mrTRG 1&2) - deferral of surgery (watch & wait) offered. 'Poor response' (mrTRG 3-5) - local colorectal MDT is informed and uses information to discuss and agree next steps in treatment and surveillance.
  Interventions: Diagnostic Test: High resolution MRI scan; Diagnostic Test: mrTRG assessment

INTERVENTIONS:
Diagnostic Test: High resolution MRI scan — MRI reporting of tumour but not mrTRG in the control arm = standard of care
Diagnostic Test: mrTRG assessment — Watch and wait offered for good responders Consider further treatment for poor responders
  Arms: Intervention arm

SUMMARY:
Open to patients undergoing any pre-operative treatment for locally advanced rectal cancer, TRIGGER is the only phase III clinical trial in the UK offering watch and wait. All patients will have post treatment MRI scans routinely performed, no change from the MERCURY trials high resolution MRI protocol is required. Patients will be randomised to either the control arm for management according to national guidelines - conventional MDT, clinical assessment post-treatment planning using the baseline MRI. Patients in the interventional arm will have their post treatment MRI scans read by a radiologist trained and supported to reliably report the mrTRG grade and have their management directed accordingly - 'Good response' (mrTRG 1&2) - watch and wait (avoidance of surgery) offered. 'Poor response' (mrTRG 3-5) - local colorectal MDT is informed and uses information to discuss and agree next steps in treatment and surveillance. Patients are followed up for five years with QoL questionnaires completed at registration, 3 and 5 years.

DETAILED DESCRIPTION:
The only phase III clinical trial in the UK offering watch and wait, the TRIGGER trial aims to validate mrTRG as an imaging biomarker for the stratified management of patients with locally advanced rectal cancer. The 'good responders' (mrTRG1&2) often have no evidence of tumour and it may be possible to avoid surgery in this group and so maintaining QoL while not impacting survival rates. The 'poor responders' (mrTRG3-5) are at high risk of poor oncological outcomes and this knowledge is useful in planning ongoing treatment and surveillance.

TRIGGER is now a non-cTIMP trial as the protocol does not specify chemotherapy or IMP treatments. Decisions about the use of chemotherapy will be based upon local MDT discussions as is normal practice and national policy and the trial CRFs will capture these decisions and whether more treatment is given to patients or not. TRIGGER does not mandate or recommend the use of any treatments: specifically it does not suggest the use of investigational medicinal products. If any centre wishes to use IMPs this would be in the context of separate trial protocols and would not preclude entry into TRIGGER.

ELIGIBILITY:
Inclusion Criteria:

1. MRI defined locally advanced rectal carcinoma i.e. one or more: greater than or equal to mrT3c; mrEMVI positive; mr N1c; mr CRM positive
2. Biopsy confirmed adenocarcinoma of radiologically defined rectum
3. Be deemed to require preoperative chemoradiotherapy (CRT) or total neoadjuvant therapy (TNT)

Exclusion Criteria:

1. Metastatic disease
2. MRI, radiotherapy and/or chemotherapy contraindications
3. A post-treatment MRI performed more than 10 weeks after the completion of radiotherapy if given
4. Previous malignancy within preceding 5 years if risk of recurrence >5%

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 441 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
To show that patients can successfully avoid surgery after achieving a good response to treatment as measured on MRI (mrTRG). | Up to 5 years
  Non-inferiority of overall survival at 3 years for the mrTRG (MRI Tumour Regression Grade) good response group (mrTRG 1 and 2) compared with control.

SECONDARY OUTCOMES:
To describe the prognostic features associated with good and poor response to treatment as measured by MRI (mrTRG) | 3 years and 5 years
  Correlation of baseline and post treatment prognostic factors on imaging and pathology against survival outcomes
To show mrTRG (Tumour Regression Grade) as a measurement tool can be reproduced by appropriately trained radiologists. | Up to 2 years
  Agreement between local and centrally measured mrTRG (MRI Tumour Regression Grade) (mrTRG 1 good to mrTRG 5 poor)
Surgical morbidity | 30 days post operative
  Comparison by arm of early (30 day) surgical morbidity according to the Clavien-Dindo classification.
Surgical morbidity | 12 months post operative
  Comparison by arm of late (up to 12 months) surgical morbidity according to the Clavien-Dindo classification.
To investigate the effect of the preoperative treatment regime on mrTRG measurement | Up to 2 years, 3 years and 5 years
  Reporting of treatment given against measurement of mrTRG (MRI Tumour Regression Grade) response (mrTRG 1 good to mrTRG 5 poor)
To investigate the effect of the preoperative treatment regime on survival outcomes | Up to 2 years, 3 years and 5 years
  Reporting of treatment given survival outcomes
To investigate the effect of mrTRG directed treatment strategy on Quality of Life | 1 year, 2 years, 3 years and 5 years
  Quality of life assessed using EORTC QLQ-C30, EQ-5D and Low Anterior Resection Syndrome Score (LARS).scans performed at baseline, post-CRT and during surveillance schedule.
To investigate the economic impact of introducing an mrTRG directed treatment strategy | Up to 2 years, 3 years and 5 years
  Healthcare costs using NHS Reference Costs combined with health resource utilization and QoL data
To define molecular and immunological characteristics associated with treatment response as measured by MRI (mrTRG). | Up to 2 years, 3 years and 5 years
  Correlate molecular and immunological biomarkers with outcome measures of mrTRG (MRI Tumour Regression Grade) response, (mrTRG 1 good to mrTRG 5 poor) and survival outcomes
To assess whether the detection of ctDNA predicts for relapse in patients with locally advanced rectal cancer | Up to 2 years, 3 years and 5 years
  Correlate ctDNA levels with outcome measures of mrTRG (MRI Tumour Regression Grade) (mrTRG 1 good to mrTRG 5 poor) and survival outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (10):
- United Kingdom (10):
  - Aberdeen Royal Infirmary - NHS Grampion, Aberdeen, Aberdeenshire
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - University Hospital of North Midlands NHS Trust - Royal Stoke, Stoke-on-Trent, Staffordshire
  - Salisbury NHS Foundation Trust, Salisbury, Wiltshire
  - Bristol Royal Infirmary, Bristol
  - Colchester General Hospital, Colchester
  - NHS Lanarkshire - Hairmyres Hospital, East Kilbride
  - Diana Princess of Wales Hospital, Grimsby
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Battersby NJ, Dattani M, Rao S, Cunningham D, Tait D, Adams R, Moran BJ, Khakoo S, Tekkis P, Rasheed S, Mirnezami A, Quirke P, West NP, Nagtegaal I, Chong I, Sadanandam A, Valeri N, Thomas K, Frost M, Brown G. A rectal cancer feasibility study with an embedded phase III trial design assessing magnetic resonance tumour regression grade (mrTRG) as a novel biomarker to stratify management by good and poor response to chemoradiotherapy (TRIGGER): study protocol for a randomised controlled trial. Trials. 2017 Aug 29;18(1):394. doi: 10.1186/s13063-017-2085-2. PMID 28851403